CLINICAL TRIAL: NCT06677918
Title: A Randomised, Double-blind, Placebo-controlled Trial to Assess the Effects of EP395 Following an Inhaled Endotoxin Challenge in Healthy Adults
Brief Title: Clinical Trial Investigating the Effects of EP395 Following an Inhaled Endotoxin Challenge in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpiEndo Pharmaceuticals (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EP395-006; 2024-516187-29-00 (EU CTIS Number); U1111-1310-4490 (Other: WHO UTN Number)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: During the study, study participants, investigators, the sponsor, and all other persons involved in the conduct of the study will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP395 (Experimental): EP395 repeated doses (oral administration). Cohort A: daily (1 capsule) for 21 days. Cohort B (optional): every other day (1 capsule) for 21 days
  Interventions: Drug: EP395
- Placebo (Placebo Comparator): Matched placebo capsule (oral administration). Cohort A: daily (1 capsule) for 21 days. Cohort B (optional): every other day (1 capsule) for 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EP395 — Capsule for oral use
  Arms: EP395
Drug: Placebo — Capsule for oral use
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to assess the effect of EP395 in a model of lung inflammation (inhaled lipopolysaccharide, which causes temporary inflammation in the airways). In addition, further information on the safety and tolerability of EP395 will be collected.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial in healthy adults. The study will assess the effect of repeated doses of EP395 on blood and lung markers of inflammation after inhaled lipopolysaccharide (LPS). It will also assess the safety, tolerability and systemic exposure of EP395.

Participants will be randomized to receive EP395 or placebo (taken orally) for 21 days. On Day 21, participants will inhale LPS to induce airway inflammation. Blood and sputum (phlegm) samples will be taken before and after the LPS challenge to measure inflammatory markers. A final safety follow-up visit will be performed on Day 37.

Depending on the results from the first cohort of participants (Cohort A), a second cohort may be recruited to test a lower dose of EP395 (Cohort B).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand the requirements and restrictions of the study, and to provide voluntary, written informed consent.
2. Aged ≥18 and ≤55 years at the time of signing the consent form.
3. Body mass index (BMI) of ≥19.0 and ≤31.0 kg/m^2 at Screening.
4. Medically healthy without abnormal clinically significant medical history, physical findings, vital signs, ECG and laboratory values at the time of Screening, as judged by the investigator.
5. Non-smoker, or former smoker with less than 10 pack years who stopped smoking (including e-cigarettes) at least 6 months before Screening.
6. Normal pulmonary function test (spirometry) adjusted for sex, height, and age.
7. Women of childbearing potential (WOCBP) must have a negative pregnancy test at Screening (blood) and Day 1 (urine) and must agree to use, highly effective measures of contraceptive control during trial participation and until 90 days after the last intake of study drug.

Women defined as of non-childbearing potential are postmenopausal (no menses for at least 1 year without alternative medical cause or surgically sterile women (tubal ligation, hysterectomy, or bilateral oophorectomy).

Men must agree to use a condom during sexual intercourse with WOCBP during treatment and for 90 days after the last IMP intake and should not donate sperm during this time.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the trial, or influence the results, or the participant's ability to participate in the trial.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study drug.
3. Recent infection, including but not limited to SARS-CoV-2, within 14 days prior to the sputum screening collection or Day 1.
4. Presence or history of lung disease, e.g., asthma or COPD.
5. History of or active tuberculosis at the time of Screening based on participant anamnesis. Participants who have been living together with another person with active tuberculosis at any time over the past 10 years will also be excluded.
6. Clinically significant abnormality on 12-lead ECG at Screening or Day 1 pre-dose.
7. Abnormal renal function at Screening.
8. Elevated liver values of Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 1.5 x upper limit of normal at Screening.
9. Use of prescription or non-prescription medications or herbal remedies within 28 days prior to Day 1, or unable to refrain from prescription or non-prescription medications or herbal remedies during the trial, with the exception of hormone replacement therapy, contraception and occasional use of paracetamol.
10. Live vaccine within 28 days or any other vaccine within 14 days prior to Day 1 until 28 days after the final dose.
11. Any positive result at Screening for serum hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
12. Positive drugs of abuse, smoking, or alcohol test at Screening or Day 1.
13. History of alcohol abuse or excessive intake of alcohol, as judged by the investigator.
14. Presence or history of drug abuse, as judged by the investigator.
15. Pregnant, currently breastfeeding, or intend to become pregnant during the course of the trial.
16. Known hypersensitivity to LPS, macrolides or EP395 or any of the study products.
17. Any clinically significant allergy, as judged by the investigator.
18. Planned treatment or treatment with another investigational drug within 5 half-lives or 3 months before the first administration of study drug, whichever is longer. Participants consented and screened, but not dosed in a previous clinical trial are not excluded.
19. Blood donation (or corresponding blood loss) greater than 400 mL, during the 3 months before the first administration of study drug.
20. Employees of the sponsor or employees or relatives of the investigator.
21. The investigator considers the participant unlikely to comply with trial procedures, restrictions and requirements.
22. Withdrawal of consent before randomisation (despite meeting the other eligibility criteria).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Blood surfactant protein-D (SP-D) | Day 21
  Change from baseline (pre-LPS) in blood SP-D on Day 21.

SECONDARY OUTCOMES:
Blood biomarkers of immune response and systemic inflammation | Day 21
  Change from baseline (pre-LPS) in blood biomarkers on Day 21.
Lung inflammatory markers in exhaled particles (PEx) | Day 21
  Change from baseline (pre-LPS) in PEx biomarkers on Day 21.
Plasma levels of EP395 | Day 1, 7, 13, 21 and 22
Assessment of adverse event (AE) occurrence | Day 1 to Day 37
Electrocardiogram (ECG) recording | Screening, Day 1, 7, 13, 21, 22 and 37
  12-lead ECG recording to determine ventricular rate, ECG heart rate, RR interval, PR interval, QRS duration, QT interval (uncorrected), and QT interval corrected by Fredericia's formula (QTcF).
  Absolute values and changes from baseline will be summarized for all assessed time points.
Assessment of laboratory values (haematology) | Screening, Day 1, 7, 13, 21, and 37
  Absolute values and changes from baseline will be summarized for all assessed time points .
Assessment of laboratory values (blood biochemistry) | Screening, Day 1, 7, 13, 21, and 37
  Absolute values and changes from baseline will be summarized for all assessed time points.
Vital signs - Heart rate | Screening, Day 1, 7, 13, 21, and 37
  Absolute values and changes from baseline will be summarized for all assessed time points.
Vital signs: Systolic and diastolic blood pressure | Screening, Day 1, 7, 13, 21, and 37
  Absolute values and changes from baseline will be summarized for all assessed time points.
Vital signs - Body temperature | Screening, Day 1, 7, 13, 21, and 37
  Absolute values and changes from baseline will be summarized for all assessed time points.
Physical Examination | Screening, Day 1, 13, 21, and 37
  Standard routine physical examination. Clinically significant changes will be reported as AEs.

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer Institute for Toxicology and Experimental Medicine ITEM, Division of Clinical Airway Research, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No